CLINICAL TRIAL: NCT06844032
Title: Clinical, Hemodynamic and Neurohumoral Predictors of Poor Prognosis in Heart Failure with Preserved Ejection Fraction
Brief Title: Predictors of Poor Prognosis in HFpEF
Status: Recruiting | Type: Observational
Sponsor: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Responsible Party: Principal Investigator, Anastasiia Filatova, MD, PhD, principal investigator, MD, National Medical Research Center for Cardiology, Ministry of Health of Russian Federation
Other Study IDs: AAAA-A18-118022290061-03
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: HFpEF
Keywords: HFpEF; HF; diastolic dysfunction; left ventricle (LV) filling pressures; left ventricular hypertrophy; cardiac reserves; myocardial fibrosis
MeSH Terms: conditions — Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- with primary outcome: Patients with HFpEF who experienced primary outcome (were hospitalized for HF or died)
- without primary outcome: Patients with HFpEF who survived without hospitalization for HF

SUMMARY:
Patients with HFpEF who have undergone meticulous clinical and instrumental evaluation (including diastolic exercise testing) between 2013 and 2020, will be followed up for at least 3 years.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) is a serious condition with an unfavorable prognosis.

The investigators aimed to evaluate in patients with HFpEF:

* the prognostic significance of standard resting hemodynamic parameters compared to key cardiac reserves;
* the prognostic significance of clinical parameters (sex, age, NYHA class, extra-cardiac diseases, therapy);
* the prognostic significance of biological markers of hemodynamic stress and biomarkers of inflammation and fibrosis;
* to identify independent predictors of adverse prognosis of HFpEF.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and data informed consent;
2. New York Heart Association (NYHA) class II-III heart failure;
3. Left ventricular ejection fraction > 50%;
4. Elevated LV filling pressures assessed by echocardiography at rest or at peak exercise.

Exclusion Criteria:

1. Evidence of myocardial ischemia during stress echocardiography;
2. Significant lesions of the main coronary arteries;
3. Genetic forms of HFpEF (HCM, amyloidosis, Fabry disease, glycogen storage diseases etc.);
4. Peripartum cardiomyopathy, chemotherapy-induced cardiomyopathy, viral myocarditis, isolated right-sided HF without left-sided structural disease, constrictive pericarditis, significant pericardial effusion;
5. Significant lung disease (severe lung disease requiring home oxygen or chronic oral steroid therapy);
6. Primary pulmonary artery hypertension;
7. Significant left-sided structural valve disease;
8. Anemia (Hb < 100 g/L);
9. Impaired renal function, defined as estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 (CKD-EPI);
10. Non-cardiac conditions that complicate/exclude participation in the study;
11. Exacerbation of heart failure less than 3 months prior to study entry.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with HFpEF who underwent meticulous clinical evaluation between 2013 and 2020 at the National Medical Research Centre for Cardiology (Moscow, Russian Federation)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospitalization for exacerbation of HF | From enrollment to August 2025
All-cause mortality | From enrollment to August 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budgetary Institution NATIONAL MEDICAL RESEARCH CENTRE OF CARDIOLOGY NAMED AFTER ACADEMICIAN E.I.CHAZOV. of the Ministry of Health of the Russian Federation, Moscow, Russia